CLINICAL TRIAL: NCT00306241
Title: A Phase III, Double-blind, Randomized, Controlled Study to Evaluate Immunogenicity and Safety of GSK Biologicals' HPV-16/18 L1 VLP AS04 Vaccine, Administered Intramuscularly (0, 1, 6 Month Schedule) in Healthy Females Aged 18 - 35 Years
Brief Title: A Study to Evaluate the Immunogenicity and Safety of GSK Biologicals' HPV Vaccine in Healthy Women Aged 18-35 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 106001
Record Dates: First submitted 2006-03-16; First posted 2006-03-23 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: Cervical neoplasia; Cervical cancer; Double-blind; HPV-16/18 L1 VLP AS04; HPV; AS04
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Biological: HPV-16/18 L1 VLP AS04

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. Indeed, the infection of the cervix by certain oncogenic types of HPV, if not cleared , can lead over time to cervical cancer in women . This study will evaluate the immune response induced by the HPV-16/18 L1 VLP AS04 vaccine and the safety of the vaccine.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The protocol was primarily amended for the following reason:

Merck's tetravalent HPV vaccine, Gardasil®, has been licensed and is now becoming commercially available in an increasing number of countries. Therefore, the study procedures were revised to include questions at every visit to determine if subjects have received an HPV vaccine outside of the study.

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A female of Chinese origin, residing in Hong Kong aged between, and including, 18 and 35 years at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry must be abstinent or must be using adequate contraceptive precautions for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study/ control vaccine within 30 days preceding the first dose of study/ control vaccine, or planned use during the study period.
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study/ control vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within three months preceding the first dose of study/ control vaccine or planned administration during the study period. Enrolment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates to HPV-16 and HPV-18 as assessed by enzyme-linked immunosorbent assay (ELISA) | At Month 7

SECONDARY OUTCOMES:
Occurrence of SAEs | Throughout the study period (up to Month 7)
Occurrence, intensity and relationship to vaccination of solicited general symptoms, and occurrence and intensity of solicited local symptoms | During the 7 days after each and any vaccination
Occurrence, intensity and causal relationship to vaccination of unsolicited symptoms | Within 30 days after any vaccination
Occurrence of new onset chronic diseases and other medically significant conditions regardless of causal relationship to vaccination and intensity. | Throughout the study period (up to Month 7)
Anti-HPV-16/18 antibody titres (by ELISA) | At Month 0 and Month 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ngan HY, Cheung AN, Tam KF, Chan KK, Tang HW, Bi D, Descamps D, Bock HL. Human papillomavirus-16/18 AS04-adjuvanted cervical cancer vaccine: immunogenicity and safety in healthy Chinese women from Hong Kong. Hong Kong Med J. 2010 Jun;16(3):171-9. PMID 20519752
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register